CLINICAL TRIAL: NCT04076241
Title: Effects of Adding Yoga Respiratory Training to Osteopathic Manipulative Treatment on Exhaled Nitric Oxide Level and Cardiopulmonary Function in Patients With Pulmonary Arterial Hypertension
Brief Title: Effects of Adding Yoga Respiratory Training to Osteopathic Manipulative Treatment in Pulmonary Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Baha Naci, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/0180
Record Dates: First submitted 2019-08-28; First posted 2019-09-03 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary arterial hypertension; Yoga respiratory training; Osteopathic manipulative treatment; Exhaled nitric oxide; Cardiopulmonary function
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined intervention (Experimental): Combined intervention group consisted of 16 pulmonary arterial hypertension (PAH) patients. Three different yoga breathing exercises were applied after osteopathic manipulative treatment (OMT). This combined intervention was applied 2 times a week for a period of 8 weeks with a total of 16 training sessions. There remained a 3-workday gap between two sessions. Patients in this group were thought about pathophysiology of PAH, benefits of physical activity, airway clearance, oxygen therapy, and importance of proper nutrition, adequate sleep, effective breathing after baseline assessment.
  Interventions: Other: Osteopathic manipulative treatment; Other: Yoga respiratory training
- Osteopathic manipulative treatment (Active Comparator): OMT group consisted of 16 PAH patients. Six different OMT techniques were applied 2 times a week for a period of 8 weeks with a total of 16 sessions. The same osteopathic manipulative treatment techniques applied to combined intervention group were used for this study group. There remained a 3-workday gap between two sessions. Patients in this group were thought about pathophysiology of PAH, benefits of physical activity, airway clearance, oxygen therapy, and importance of proper nutrition, adequate sleep, effective breathing after baseline assessment.
  Interventions: Other: Osteopathic manipulative treatment
- Control (No Intervention): Control group also consisted of 16 PAH patients and serves as the controls. No interventions were applied for the patients in this group. Similar with the patients in other two groups, pharmacological treatment of the patients in this group continued and they were advised for using their medication properly, Patients in this group were also thought about pathophysiology of PAH, benefits of physical activity, airway clearance, oxygen therapy, and importance of proper nutrition, adequate sleep, effective breathing after baseline assessment.

INTERVENTIONS:
Other: Osteopathic manipulative treatment — The investigators applied six different OMT techniques including rib raising, diaphragm release, suboccipital decompression, first rib mobilization, mediastinum mobilization and thoracic inlet myofascial release. Rib raising is used to increase the mobility of the rib cage and to reduce vasoconstriction by regulating sympathetic tone. Diaphragm release is used to increase diaphragm movement. Suboccipital decompression involves traction of the base of the skull. We aim to improve respiration with mobilization of the first rib which is associated with sternum, sympathetic truncus and important vascular structures. Thoracic inlet is an important structure resisting intrathoracic pressure changes during respiration. Finally, the goal of the mediastinum mobilization is to increase the mobility of the rib cage by providing relaxation in the tension of the facial tissues.
  Arms: Combined intervention; Osteopathic manipulative treatment
Other: Yoga respiratory training — Nadishodhana pranayama (Alternate nostril breathing), Ujjayi pranayama (Psychic breath) and Bhramari pranayama (Humming bee breath) were used for the study. Nadishodhana is one of the most common yoga breathing exercises and involves breathing through one nostril while closing the other one. The patients performed 2 sets of 8 breathing cycles with a resting time of 2 minutes between the sets. Ujjayi Pranayama involves soft contraction of laryngeal muscles and the partial closure of the glottis. The patients performed 2 sets of 10 breathing cycles per session with an inspiration:expiration phase as 1:2. Bhramari Pranayama includes a nasal humming sound during exhalation to create slight vibrations on the laryngeal walls, and the inner walls of the nostrils. The patients applied 2 sets of 10 breathing cycles per session with a respiration rate of 3-4/min.
  Arms: Combined intervention

SUMMARY:
The investigators planned a randomized controlled study to investigate the effects of adding yoga respiratory training to osteopathic manipulative treatment (OMT), and OMT alone on exhaled nitric oxide level and cardiopulmonary function in patients with pulmonary arterial hypertension (PAH). Our hypothesis is that combined intervention including OMT and yoga respiratory training may improve exhaled nitric oxide level and cardiopulmonary function in patients with PAH.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is characterized by a mean pulmonary arterial pressure of >20 mmHg, measured by right heart catheterization at rest. PAH begins in the small arteries of the pulmonary vasculature and is characterized by increased vasoconstriction. Pulmonary vasodilatation induced by perivascular nerve stimulation usually occurs with nitric oxide (NO). A decrease in the airway wall concentration of NO was detected in patients with PAH. It has been reported that patients with PAH have a mild to moderate decrease in lung volumes associated with disease severity. A decrease in exercise capacity and respiratory muscle strength has been reported in patients with PAH.

Osteopathic Manipulative Therapy (OMT) is a well-known manual therapy approved by World Health Organization. A single-session of OMT was found to increase pulmonary function, inspiratory muscle strength, oxygen saturation, and to reduce dyspnea and fatigue in individuals with severe chronic obstructive pulmonary disease. It has been observed that OMT increases parasympathetic activity and reduces blood pressure in patients with hypertension.

Pranayama breathing is an important component of of yoga. It has been reported that yoga respiratory training increases vagal tone and reduces sympathetic activity, increases vital capacity, controls heart rate and blood pressure, and improves respiratory muscle strength.

No study investigating the effects of adding yoga respiratory training to osteopathic manipulative treatment in patients with PAH was found in the literature. The investigators aimed to explore the effects of a combined intervention consisting of OMT and yoga breathing exercises, as well as OMT alone on exhaled NO level, pulmonary function, respiratory and peripheral muscle strength, and exercise capacity in patients with PAH.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary hypertension patients that are clinically and hemodynamically stable
* Resting mean pulmonary arterial pressure > 20 millimeter of mercury (mmHg) during a right heart catheterization
* Being over 18 years old
* Volunteering to participate in the study and to sign a written informed consent form
* Patients with New York Heart Association (NYHA) functional class I-II-III
* Stable pulmonary hypertension patients that takes medication at least 3 months.

Exclusion Criteria:

* Acute decompensated heart failure
* Unstable angina pectoris
* Recent thoracic or abdominal surgical procedures
* Severe neurological impairments
* Severe cognitive impairment
* Recent syncope
* Using the immune system drugs as a result of organ or tissue transplants
* Fractures within the past six months
* Osteoporosis
* Tumors
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-09-07 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Forced Vital Capacity (FVC), Forced Expiratory Volume in One Second (FEV1) at 8 weeks | Baseline and week 8
  FVC and FEV1 were recorded in liter (l) by using spirometry (Spiro USB, CareFusion US). Measurements were performed according to American Thoracic Society/European Respiratory Society (ATS/ERS) recommendations.
Change from Baseline Forced Expiratory Volume in One Second/Forced Vital Capacity (FEV1/FVC) at 8 weeks | Baseline and week 8
  FEV1/FVC ratio (%) was recorded with regards to the highest FEV1 and FVC values measured by spirometry.
Change from Baseline Forced Expiratory Flow at 25-75% of FVC (FEF25-75) at 8 weeks | Baseline and week 8
  FEF25-75 was recorded in liter/second (l/s) by using spirometry (Spiro USB, CareFusion US). Measurements were performed according to American Thoracic Society/European Respiratory Society (ATS/ERS) recommendations.
Change from Baseline Peak Expiratory Flow (PEF) at 8 weeks | Baseline and week 8
  PEF was recorded in liter/minute (l/min) by using spirometry (Spiro USB, CareFusion US). Measurements were performed according to American Thoracic Society/European Respiratory Society (ATS/ERS) recommendations.
Change from Baseline FVC%, FEV1%, FEF25-75%, PEF% at 8 weeks | Baseline and week 8
  FVC%, FEV1%, FEF25-75% and PEF% were recorded as the percentage of predicted values.
Change from Baseline Nitric Oxide Level at 8 weeks | Baseline and week 8
  Fractional Exhaled Nitric Oxide (FeNO) was measured according to ATS/ERS recommendations with a hand-held, portable device (NObreath, Bedfont, UK). After inhaling the ambient air for 2-3 seconds until the total lung capacity, the patient is asked to exhale into the device for more than 6 seconds at constant flow rate (50 milliliter/second) without holding breath. The mean of two technically acceptable values within 10% was recorded in parts per billion (ppb) and maximum six attempts were performed.
Change from Baseline Exercise Capacity at 8 weeks | Baseline and week 8
  Exercise capacity was measured with the 6 Minute Walk Test (6MWT) according to the ATS guidelines. The 6 minutes wallking distance (6MWD) was recorded in meters. Higher scores indicate a better outcome.
Change from Baseline 6MWD% at 8 weeks | Baseline and week 8
  6MWD% was recorded as the percentage of predicted distances. Higher scores indicate a better outcome.
Change from Baseline Changes of Perceived Dyspnea and Fatigue at 8 weeks | Baseline and week 8
  Perceived dyspnea and fatigue were measured before and immediately after 6MWT with modified Borg scale ranging from 0 to 10. Higher scores indicate a worse outcome. Changes of perceived dyspnea and fatigue were recorded.
Change from Baseline Resting Peripheral Oxygen Saturation (SpO2) at 8 weeks | Baseline and week 8
  SpO2 was measured by using a pulse oximeter and was recorded as percentage.
Change from Baseline Change of Blood Pressure at 8 weeks | Baseline and week 8
  Systolic and diastolic blood pressures were measured before and immediately after 6MWT with sphygmomanometer. Change of systolic blood pressure and change of diastolic blood pressure were recorded.
Change from Baseline Resting Heart Rate at 8 weeks | Baseline and week 8
  Resting heart rate was measured with a pulse oximeter and was recorded as beats per minute (bpm).

SECONDARY OUTCOMES:
Change from Baseline Respiratory Muscle Strength at 8 weeks | Baseline and week 8
  MIP and MEP were recorded as cmH2O, as well as MIP% and MEP% were recorded as the percentage of predicted values according to age and gender, as described by Black and Hyatt.
Change from Baseline Peripheral Muscle Strength at 8 weeks | Baseline and week 8
  Hand grip strength was measured with a hand-held dynamometer bilaterally. Three measurements on both hands were performed and the highest values were recorded in kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: Baha Naci, PhD., Principal Investigator — Istanbul University - Cerrahpasa; Rengin Demir, PhD., Study Director — Istanbul University - Cerrahpasa; Mehmet Serdar Kucukoglu, MD, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Cardiology Institute, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M; ESC Scientific Document Group. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Heart J. 2016 Jan 1;37(1):67-119. doi: 10.1093/eurheartj/ehv317. Epub 2015 Aug 29. No abstract available. PMID 26320113
- [Background] McLaughlin VV, Archer SL, Badesch DB, Barst RJ, Farber HW, Lindner JR, Mathier MA, McGoon MD, Park MH, Rosenson RS, Rubin LJ, Tapson VF, Varga J, Harrington RA, Anderson JL, Bates ER, Bridges CR, Eisenberg MJ, Ferrari VA, Grines CL, Hlatky MA, Jacobs AK, Kaul S, Lichtenberg RC, Lindner JR, Moliterno DJ, Mukherjee D, Pohost GM, Rosenson RS, Schofield RS, Shubrooks SJ, Stein JH, Tracy CM, Weitz HH, Wesley DJ; ACCF/AHA. ACCF/AHA 2009 expert consensus document on pulmonary hypertension: a report of the American College of Cardiology Foundation Task Force on Expert Consensus Documents and the American Heart Association: developed in collaboration with the American College of Chest Physicians, American Thoracic Society, Inc., and the Pulmonary Hypertension Association. Circulation. 2009 Apr 28;119(16):2250-94. doi: 10.1161/CIRCULATIONAHA.109.192230. Epub 2009 Mar 30. No abstract available. PMID 19332472
- [Background] Ayajiki K, Okamura T, Noda K, Toda N. Functional study on nitroxidergic nerve in isolated dog pulmonary arteries and veins. Jpn J Pharmacol. 2002 Jun;89(2):197-200. doi: 10.1254/jjp.89.197. PMID 12120765
- [Background] World Health Organization (WHO) Benchmarks for training in traditional/complementary and alternative medicine: benchmarks for training in osteopathy. Geneva: WHO Press; 2010.
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Black LF, Hyatt RE. Maximal respiratory pressures: normal values and relationship to age and sex. Am Rev Respir Dis. 1969 May;99(5):696-702. doi: 10.1164/arrd.1969.99.5.696. No abstract available. PMID 5772056
- [Background] American Thoracic Society; European Respiratory Society. ATS/ERS recommendations for standardized procedures for the online and offline measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide, 2005. Am J Respir Crit Care Med. 2005 Apr 15;171(8):912-30. doi: 10.1164/rccm.200406-710ST. No abstract available. PMID 15817806
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Result] Girgis RE, Champion HC, Diette GB, Johns RA, Permutt S, Sylvester JT. Decreased exhaled nitric oxide in pulmonary arterial hypertension: response to bosentan therapy. Am J Respir Crit Care Med. 2005 Aug 1;172(3):352-7. doi: 10.1164/rccm.200412-1684OC. Epub 2005 May 5. PMID 15879413
- [Result] Sun XG, Hansen JE, Oudiz RJ, Wasserman K. Pulmonary function in primary pulmonary hypertension. J Am Coll Cardiol. 2003 Mar 19;41(6):1028-35. doi: 10.1016/s0735-1097(02)02964-9. PMID 12651053
- [Result] Desai SA, Channick RN. Exercise in patients with pulmonary arterial hypertension. J Cardiopulm Rehabil Prev. 2008 Jan-Feb;28(1):12-6. doi: 10.1097/01.HCR.0000311502.57022.73. PMID 18277824
- [Result] Kabitz HJ, Bremer HC, Schwoerer A, Sonntag F, Walterspacher S, Walker DJ, Ehlken N, Staehler G, Windisch W, Grunig E. The combination of exercise and respiratory training improves respiratory muscle function in pulmonary hypertension. Lung. 2014 Apr;192(2):321-8. doi: 10.1007/s00408-013-9542-9. Epub 2013 Dec 13. PMID 24338088
- [Result] Mereles D, Ehlken N, Kreuscher S, Ghofrani S, Hoeper MM, Halank M, Meyer FJ, Karger G, Buss J, Juenger J, Holzapfel N, Opitz C, Winkler J, Herth FF, Wilkens H, Katus HA, Olschewski H, Grunig E. Exercise and respiratory training improve exercise capacity and quality of life in patients with severe chronic pulmonary hypertension. Circulation. 2006 Oct 3;114(14):1482-9. doi: 10.1161/CIRCULATIONAHA.106.618397. Epub 2006 Sep 18. PMID 16982941
- [Result] Yilmaz Yelvar GD, Cirak Y, Demir YP, Dalkilinc M, Bozkurt B. Immediate effect of manual therapy on respiratory functions and inspiratory muscle strength in patients with COPD. Int J Chron Obstruct Pulmon Dis. 2016 Jun 20;11:1353-7. doi: 10.2147/COPD.S107408. eCollection 2016. PMID 27382271
- [Result] Curi ACC, Maior Alves AS, Silva JG. Cardiac autonomic response after cranial technique of the fourth ventricle (cv4) compression in systemic hypertensive subjects. J Bodyw Mov Ther. 2018 Jul;22(3):666-672. doi: 10.1016/j.jbmt.2017.11.013. Epub 2017 Dec 9. PMID 30100295
- [Result] Nayar HS, Mathur RM, Kumar RS. Effects of yogic exercises on human physical efficiency. Indian J Med Res. 1975 Oct;63(10):1369-76. No abstract available. PMID 1222951
- [Result] Singh S, Gaurav V, Parkash V. Effects of a 6-week nadi-shodhana pranayama training on cardio-pulmonary parameters. J. Phys. Educ. Sport Manag. 2: 44-47, 2011.
- [Result] Garg S, Chandla SS. Effect of nadi shodhan pranayama on pulmonary functions. Int J Health Sci Res. 6: 192-196, 2016.